CLINICAL TRIAL: NCT00967083
Title: Support Needs and Preferences of Family Caregivers of Lung Cancer Patients
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Queens Cancer Center of Queens Hospital (Other); Michigan State University (Other); National Cancer Institute (NCI) (NIH); Indiana University (Other)
Responsible Party: Sponsor
Other Study IDs: 09-104
Record Dates: First submitted 2009-08-26; First posted 2009-08-27 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Lung Cancer
Keywords: Quality of Life; Questionnaires; Interviews; family members; care givers; 09-104
MeSH Terms: conditions — Lung Neoplasms | interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- family caregivers of lung cancer patients: In this 2-year pilot study, we plan to screen family caregivers of lung cancer patients within 4 to 6 weeks after the a new visit to the thoracic clinic. We will screen spouses, adult children, and other family members using the HAD-18 to determine their level of anxiety and depressive symptoms at enrollment.
  Interventions: Behavioral: Questionnaires/Interviews

INTERVENTIONS:
Behavioral: Questionnaires/Interviews — Baseline assessment of distressed caregivers within 4-6 weeks a new visit to the thoracic clinic. Three-month follow-up assessment of caregivers. Qualitative phone interviews with a subsample of 30 caregivers within 3 weeks of follow-up.

SUMMARY:
This study is being done to learn what the needs are in relation to the family members. Some family members seek counseling; others do not. The institution wants to try to understand why and wants to see if they can improve our support services for family members.

ELIGIBILITY:
Inclusion Criteria:

* Primary family caregiver identified by a patient who is approximately within 4 to 6 weeks of a new visit to a thoracic clinic and receiving cancer care at Memorial Sloan-Kettering Cancer Center or Queens Cancer Center
* Caregiver is at least 18 years of age.
* Caregiver has adequate English fluency for completion of data collection. The surveys were designed and validated in English and are not currently available in other languages. Translation of questionnaires into other languages would require reestablishing the reliability and validity of these measures. Therefore, participants must be able to communicate in English to complete the surveys.
* Clinically meaningful distress defined as a score of 8 or greater on the Anxiety or Depression subscale of the HADS (see Bjelland et al., 2002; Zigmond & Snaith, 1983).

Exclusion Criteria:

* Patients or caregivers exhibiting significant psychiatric or cognitive impairment (dementia/delirium, retardation, active psychosis) that in the judgment of the investigators would preclude providing informed consent and study participation
* Patient has lung cancer recurrence
* Currently participating in a psychosocial intervention trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients whose family caregivers may be eligible for this study will be identified by a member of the patient's treatment team, the protocol investigator, or research team at Memorial Sloan-Kettering Cancer Center (MSKCC) or Queens Cancer Center (QCC).
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2009-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Assess psychosocial info & practical needs of prim family caregivers of lung cancer pts.Mental health (anxiety & depression)& behavioral health needs(smoking cessation,alcohol abuse)will be assessed b/c these 2 types of needs are strongly correlate | 13 to 16 weeks

SECONDARY OUTCOMES:
To assess psychosocial and practical barriers to psychosocial support service use among primary family caregivers of lung cancer patients | 13 to 16 weeks
To assess family caregivers' preferences (preferred topics, modality, provider, timing) regarding psychosocial support interventions. | 13 to 16 weeks
To gather descriptive information regarding participant flow for planning future intervention studies. | 13 to 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Ostroff, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Queens Cancer Center of Queens Hospital, Jamaica, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm